CLINICAL TRIAL: NCT00778115
Title: A Relative Bioavailability Study of Loperamide HCl 2 mg and Simethicone 125 mg Tablets to Imodium® Advanced Caplets Under Fasting Condition
Brief Title: Bioequivalence Study of Loperamide Hydrochloride 2 mg and Simethicone 125 mg Tablet Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: B045521
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence Loperamide HCl 2 mg and simethicone 125 mg tablets
MeSH Terms: interventions — Loperamide; Simethicone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Loperamide HCl 2 mg and simethicone 125 mg tablets of ranbaxy
  Interventions: Drug: Loperamide HCl 2 mg and simethicone 125 mg tablets
- 2 (Active Comparator): Imodium® Advanced caplets
  Interventions: Drug: Loperamide HCl 2 mg and simethicone 125 mg tablets

INTERVENTIONS:
Drug: Loperamide HCl 2 mg and simethicone 125 mg tablets

SUMMARY:
The objective of this study is to compare the relative bioavailability of Loperamide HCl 2 mg and simethicone 125 mg tablets (Ranbaxy) with that of Imodium® Advanced caplets (McNeil) in healthy subjects under fasting condition

DETAILED DESCRIPTION:
The study was conducted as a single-dose, randomized, 2-period sequence crossover study under fasting condition comparing equal dose of test and reference products with an interval period of at least 7 days. The period of confinement was at least 10 hours before dosing until after 24 hours blood collection in each period. Subjects were asked to return to the clinic for subsequent blood circulation Twenty-six subjects (26) were recruited for the study of which twenty-three (23) completed the clinical portion of the study. Subject #17 was withdrawn by sponsor's representative due to adverse event unrelated to the drug), subject #18 and subject #25 voluntarily withdrew due to adverse event

ELIGIBILITY:
Inclusion Criteria:

1. All subjects selected for this sudy will be at least 18 years of age
2. Each subjects shall be given a general physical examination within 28 days of initiation of the study. Such examination includes, but is not limited to, blood pressure, general observations, and history
3. Each female subject will be given a serum pregnancy test as part of the pre-study screening process At the end of the study, the subjects will have an exit evaluation, and clinical laboratory measurements Adequate blood and urine samples should be obtained within 28 days before beginning of the first period and at the end of the clinical laboratory measurements Clinical laboratory measurement will include the haematology, clinical chemistry, urine analysis, HIV screen, Hepatitis-B,C screen, Drugs of abuse screen

Exclusion Criteria:

Subject candidates who met the following criteria were excluded::

1. Subjects with a history of alcoholism or drug addiction (during past 2 years), or serious gastrointestinal, renal, hepatic or cardiovascular disease, tuberculosis, epilepsy, asthma, diabetes, psychosis or glaucoma will not be eligible for study
2. Subjects whose clinical laboratory tests are outside the normal range may be retested at the request of clinical investigator. If the clinical values are outside this range on retesting, subject will not be eligible to participate in the study unless the clinical investigator deems the result to not to be significant
3. Subjects who have a history of allergic responses to the class of drug being tested should be excluded from the study
4. All subjects will have urine samples assayed for the presence of drugs of abuse as a part of the clinical laboratory screening procedure and at each check-in. Subjects found to have urine concentrations of any of the tested drugs will not be allowed to participate
5. Subjects should not have donated blood and/ or plasma for at least 30 days prior to the first dosing of the study
6. Subjects who have taken investigational drug within 30 days prior to the first dosing of the study
7. Female subjects who are pregnant, breast feeding, or who are likely to become pregnant during the study will not be allowed to participate. Female subjects of child bearing potential must either abstain from sexual intercourse or use a reliable barrier method (eg. Condom, IUD) of contraception during course of the study or they will not be allowed to participate. Subjects who have used implanted or injected hormonal contraceptives before 14 days of dosing will not be allowed to participate
8. All female subjects will be screened for pregnancy at check-in in each period. Subjects with positive or inconclusive results will be withdrawn from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2004-11; Primary Completion 2004-11 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- Gateway Medical Research, Inc., Saint Charles, Missouri, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html